CLINICAL TRIAL: NCT01768637
Title: Whole Blood Platelet Aggregation in Chronic Kidney Disease Patients on Aspirin
Brief Title: Whole Blood Platelet Aggregation in Chronic Kidney Disease Patients on Aspirin Study
Acronym: WiCKDonASA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12CRP11830004
Record Dates: First submitted 2013-01-10; First posted 2013-01-15 (Estimated); Results first posted 2019-04-19 (Actual); Last update posted 2019-04-19 (Actual); Status verified 2019-01

CONDITIONS: Chronic Kidney Disease
Keywords: Chronic kidney disease; Platelet function; aspirin; antiplatelet agent
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Aspirin; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chronic Kidney Disease (Experimental): Patients with pre-dialysis stages 4-5 Chronic Kidney Disease will receive open-label aspirin 81 mg once daily for 2 weeks, then 2 weeks of aspirin 81 mg plus clopidogrel 75 mg once daily.
  Interventions: Drug: Aspirin; Drug: Clopidogrel
- Normal controls (Active Comparator): Patients without Chronic Kidney Disease will receive open-label aspirin 81 mg once daily for 2 weeks, then 2 weeks of aspirin 81 mg plus clopidogrel 75 mg once daily.
  Interventions: Drug: Aspirin; Drug: Clopidogrel

INTERVENTIONS:
Drug: Aspirin — Aspirin 81 mg by mouth daily
  Other Names: ASA
Drug: Clopidogrel — Clopidogrel 75 mg by mouth once daily
  Other Names: Plavix

SUMMARY:
Higher coronary in-stent thromboses and bleeding complications on anti-platelet agents are more common in Chronic Kidney Disease vs. non-Chronic Kidney Disease patients. Poor inhibition of platelet aggregation by anti-platelet agents predicts future cardiovascular events. Clinical practice guidelines are ambiguous about the use of these agents in Chronic Kidney Disease due to lack of controlled studies. The investigators hypothesize that patients with Chronic Kidney Disease compared with non-Chronic Kidney Disease have reduced platelet aggregation and poor platelet inhibitory response to aspirin. The aims are to 1) define the range of whole blood platelet aggregation in stages 3-5 Chronic Kidney Disease patients; 2) investigate whether patients with stages 4-5 Chronic Kidney Disease vs. non-Chronic Kidney Disease have lower platelet aggregation or impaired von Willebrand Factor activity; and 3) compare inhibition of platelet aggregation from baseline after 2 weeks of aspirin therapy and another 2 weeks of clopidogrel therapy added to aspirin in Chronic Kidney Disease vs. non-Chronic Kidney Disease patients. Accomplishing these aims will provide pilot data to power future studies of targeted anti-platelet agent treatments in Chronic Kidney Disease in order to improve cardiovascular outcomes.

DETAILED DESCRIPTION:
Patients will be consented for the study and asked to initial on the consent form to state whether they agree for the genetic testing. After signing informed consent, complete medical history and medication list will be obtained and verified with the electronic medical record. After meeting all inclusion and exclusion criteria during the screening visit, those patients on aspirin for primary prevention of cardiovascular events will be asked to stop it for 2 weeks prior to blood collection for baseline data. Normal controls will be chosen after frequency matching for decade of age, gender, diabetes mellitus and interval of body mass index (5 kg/m2). Dietary supplements (Vitamin E and fish oil) known to affect platelet function will be assessed and patients on those will be asked to discontinue these. Participants with also be asked to not eat foods known to affect platelet function (coffee, chocolate, grapes, and alcohol) 48 hours prior to sample collection on visit 1. An interviewer-administered assessment of diet and exercise with a modified 24-hour dietary recall and the Stanford 7-day Physical activity Recall will be performed to ensure dietary consistency which may affect platelet aggregability on visit 1. Blood will be drawn via venopuncture for laboratory studies (whole blood platelet aggregation, von Willebrand Factor antigen levels and activity). Participants will be administered aspirin 81 mg for 2 weeks and asked to return in 2 weeks. On visit 2, whole blood platelet aggregation will be re-measured and questionnaires filled out. Two oral swabs will be taken from those participants who consented for genetic testing and samples will be stored at Dallas Veterans Affairs Medical Center for short term until shipped to Diagnostics Laboratory for genetic testing of clopidogrel cytochrome P450 polymorphisms. All participants will be administered clopidogrel 75 mg daily on top of aspirin 81 mg for 2 weeks and asked to return in 2 weeks. On visit 3, whole blood platelet aggregation will be re-measured and questionnaires filled out. At the completion of the study, participants will be placed back on their original antiplatelet agent if applicable and referred back to the primary care provider.

ELIGIBILITY:
Inclusion Criteria:

* Male or female >21 years

Cases:

Chronic kidney disease stages 4-5, with estimated glomerular filtration rate of <30

Controls:

estimated glomerular filtration rate of >90, urinary albumin to creatinine ratio <30 and no other kidney damage

Exclusion Criteria:

* End-stage renal disease (peritoneal dialysis and hemodialysis)
* Kidney transplant or any other transplant patient
* Recent hospitalizations <3 months
* Acute coronary or cerebrovascular event in the last 12 months
* Surgery in the last 3 months
* Blood dyscrasias or active bleeding
* Gastro-intestinal bleeding in the last 6 months
* Concomitant use of other anti-platelet agent or antithrombotic drugs
* Recent treatment (<30 days) with a glycoprotein antagonist or proton pump inhibitor
* Hematocrit <25% or white blood cell count >20,000 or platelet count <50,000
* Any active malignancy or liver disease
* No current diagnosis of depression, not on any antidepressant medications,

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2014-04 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Hedayati, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
we will upload informed consent form and the study protocol.
Supporting Information: Study Protocol, ICF
Time Frame: upon completion of the study and the publication
Access Criteria: everyone

REFERENCES:
- [Result] Jain N, Li X, Adams-Huet B, Sarode R, Toto RD, Banerjee S, Hedayati SS. Differences in Whole Blood Platelet Aggregation at Baseline and in Response to Aspirin and Aspirin Plus Clopidogrel in Patients With Versus Without Chronic Kidney Disease. Am J Cardiol. 2016 Feb 15;117(4):656-663. doi: 10.1016/j.amjcard.2015.11.029. Epub 2015 Dec 7. PMID 26725101
- [Derived] Jain N, Wan F, Kothari M, Adelodun A, Ware J, Sarode R, Hedayati SS. Association of platelet function with depression and its treatment with sertraline in patients with chronic kidney disease: analysis of a randomized trial. BMC Nephrol. 2019 Oct 29;20(1):395. doi: 10.1186/s12882-019-1576-7. PMID 31664940

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from December 10, 2012 to January 31, 2014 from outpatient clinics at Parkland hospital, Dallas Veterans Affairs hospital and University of Texas Southwestern Medical Center, Dallas, TX, USA.
Pre-assignment Details: From 1,545 participants screened from outpatient clinics, 196 eligible patients were approached for enrollment, 128 refused and 48 signed consent.
Period: Overall Study
Arm/Group | Chronic Kidney Disease | Normal Controls
Started (Signed consent) | 29 | 19
Completed Visit 1 | 28 | 16
Completed Visit 2 | 26 | 13
Completed (completed visit 3) | 26 | 12
Not Completed | 3 | 7
Not completed — Lost to Follow-up | 2 | 7
Not completed — Difficult blood draw | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chronic Kidney Disease | Normal Controls | Total
Number analyzed (Participants) | 28 | 16 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (10) | 49 (11) | 51 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 8 | 20
  Male | 16 | 8 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 4 | 12
  Not Hispanic or Latino | 20 | 12 | 32
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 4 | 19
  White | 13 | 12 | 25
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 32.0 (5.5) | 29.8 (4.9) | 31.2 (5.3)
Diabetes mellitus [Count of Participants; unit: Participants] | 13 | 7 | 20
Proton pump inhibitor use [Count of Participants; unit: Participants] | 1 | 1 | 2
Beta blocker use [Count of Participants; unit: Participants] | 21 | 0 | 21
Statin use [Count of Participants; unit: Participants] | 19 | 5 | 24
Angiotensin converting enzyme inhibitor or angiotensin receptor blocker use [Count of Participants; unit: Participants] | 12 | 5 | 17
Allopurinol use [Count of Participants; unit: Participants] | 6 | 0 | 6
Baseline use of aspirin [Count of Participants; unit: Participants] | 12 | 4 | 16
estimated glomerular filtration rate (eGFR) [Mean (Standard Deviation); unit: ml/min/1.73m^2] | 17 (7) | 101 (15) | 47.2 (42.3)
Urine albumin to creatinine ratio [Median (Inter-Quartile Range); unit: mg/g] | 1282 [143 to 1848] | 5 [2.5 to 8.8] | 87 [0 to 6469]
Hemoglobin [Mean (Standard Deviation); unit: g/dl] | 11.2 (1.7) | 14.4 (1.7) | 12.5 (2.3)
Hematocrit [Mean (Standard Deviation); unit: percent of red blood cells in blood] | 33.9 (5.1) | 42.6 (4.2) | 36.9 (6.4)
Platelet count [Mean (Standard Deviation); unit: K per microL] | 232 (55) | 217 (55) | 227 (54.7)
Glycosylated hemoglobin [Mean (Standard Deviation); unit: percent of glycated hemoglobin in blood] | 6.8 (0.4) | 6.4 (0.4) | 6.4 (1.3)

OUTCOME MEASURES:

1. Primary Outcome: Whole Blood Platelet Aggregation to 0.5 Millimoles Arachidonic Acid
Description: Citrated whole blood was used to measure platelet aggregation induced by agonist (arachidonic acid at 5 mM concentration) using impedance whole blood platelet aggregometry via a Chrono-log aggregometer. Values at baseline (visit 1) was compared between groups with post treatment values (visit 2) after 2 weeks of aspirin treatment
Time Frame: 2 weeks
Measure: Median (Inter-Quartile Range); unit: ohms
Arm/Group | Chronic Kidney Disease | Normal Controls
Number analyzed (Participants) | 28 | 16
ohms
  Baseline | 21.0 [10.5 to 24.5] | 18.0 [10.0 to 20.0]
  visit 2 | 0 [0 to 0] | 0 [0 to 0]

2. Secondary Outcome: Whole Blood Platelet Aggregation to 2 µg/mL Collagen
Description: Citrated whole blood was used to measure platelet aggregation induced by agonist (collagen at 2mM concentration) using impedance whole blood platelet aggregometry via a Chrono-log aggregometer. Values at baseline (visit 1) was compared between groups with post treatment values (visit 2) after 2 weeks of aspirin treatment
Time Frame: 2 weeks
Measure: Median (Inter-Quartile Range); unit: ohms
Arm/Group | Chronic Kidney Disease | Normal Controls
Number analyzed (Participants) | 28 | 16
ohms
  Baseline | 28.5 [23.5 to 31.5] | 25.0 [20.0 to 30.0]
  visit 2 | 19.5 [16.0 to 26.0] | 19.0 [16.0 to 22.0]

3. Secondary Outcome: Whole Blood Platelet Aggregation to 20 µg/mL Adenosine Diphosphate
Description: Citrated whole blood was used to measure platelet aggregation induced by agonist (adenosine diphosphate at 20mM concentration) using impedance whole blood platelet aggregometry via a Chrono-log aggregometer. Values at baseline (visit 1) and on aspirin (visit 2) was compared between groups with post treatment values (visit 3) after 2 weeks of aspirin and clopidogrel treatment
Time Frame: 4 weeks
Measure: Mean (Inter-Quartile Range); unit: ohms
Arm/Group | Chronic Kidney Disease | Normal Controls
Number analyzed (Participants) | 28 | 16
ohms
  Baseline | 13.5 [9.5 to 16.0] | 9.0 [6.0 to 12.0]
  visit 2 | 11.0 [8.0 to 16.0] | 10.0 [8.0 to 11.0]
  visit 3 | 8.0 [1.0 to 12.0] | 3.0 [0 to 4.0]

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the period of the study visits for an average of 4 weeks.
Description: not different
Arm/Group | Chronic Kidney Disease | Normal Controls
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/16
Other Adverse Events (participants affected / at risk) | 5/28 | 9/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chronic Kidney Disease (N=28) | Normal Controls (N=16)
Brusing or nose bleed (Blood and lymphatic system disorders) | 5 (5) | 9 (9)

LIMITATIONS AND CAVEATS:
Limited by residual confounding due to small sample size and lack of randomization ex vivo measurement of platelet function which may be different from in vivo function Sub-optimal reproducibility of platelet assays

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No